CLINICAL TRIAL: NCT00777205
Title: Improving Depression Management Through Peer Support
Acronym: DIAL-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 08-325
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-11

CONDITIONS: Depression
Keywords: Peer Support; Quality of Life; Telephone
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care (Active Comparator): Patients in the enhanced usual care arm received their usual mental health care, a copy of the Depression Helpbook, and bi-weekly study mailings with depression management tips.
  Interventions: Behavioral: Enhanced Usual Care
- Telephone-based peer support (Experimental): Participants in the intervention arm received usual mental health care and biweekly study mailings. In addition, they had access to a telephone platform over which they could make free calls to their peer partner for mutual peer support over a 6-month period of time.
  Interventions: Behavioral: Telephone-based peer support; Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Telephone-based peer support — Patients received a) a peer-support manual that outlines self-management and recovery principles and provides peer discussion topics and b) access to a specialized telephone platform that permits free calls to their partners, ready access to mental health staff for back-up and advice on being effective partners, and recorded tips on depression management. They were asked to call their peer partner at least once a week for 24 weeks.
  Arms: Telephone-based peer support
Behavioral: Enhanced Usual Care — Patients received their usual mental health care plus a copy of the Depression Helpbook by Wayne Katon and bi-weekly study mailings with depression management tips.

SUMMARY:
We conducted a randomized controlled trial (RCT) that compared the effectiveness of a telephone delivered, recovery focused, peer-support intervention to enhanced usual care for VA patients with depression.

DETAILED DESCRIPTION:
Peer-support interventions have been recommended by prestigious national task forces and incorporated into the VA Comprehensive Mental Health Strategic Plan. Patients who cope with longer term depressive symptoms may benefit from these interventions.This study examines the effectiveness of a feasible, scalable mutual peer-support intervention for VA patients in depression treatment and will inform leaders who are considering implementing peer-support initiatives.

In this study, each study participant (a veteran in treatment for depression) was matched with another participating veteran and the pairs were randomized to enhanced usual care or to the telephone based peer-support intervention (DIAL-UP). All study participants received usual care plus written materials outlining depression self-management strategies, behavioral activation, and recovery.

DIAL-UP participants also received: a) a peer-support manual that outlined peer support principles and provided peer discussion topics and b) access to a specialized telephone platform that permited free calls to their partners, ready access to mental health staff for back-up and advice, and recorded tips on depression management. Patients were encouraged to call their partners at least once per week during the 6-month intervention period. Patient outcomes were assessed at 3, 6, and 12 months following enrollment.

ELIGIBILITY:
Inclusion Criteria:

* currently in treatment at Ann Arbor, Detroit, Battle Creek, or Saginaw VA or their associated community based outpatient clinics
* not receiving formal mental health services or regularly attending mutual self-help programs outside of the VA
* diagnosis of a depressive disorder in the last 24 months that is confirmed by the relevant clinician
* being seen less than bi-weekly by clinicians for psychiatric or substance use disorders
* past trial of psychotherapy and/or antidepressant trial
* have a current PHQ-9 scores > 10 or WSAS scores > 10
* have stable access to and ability to communicate by telephone

Exclusion Criteria:

* diagnosis of schizophrenia, schizoaffective disorder, MDD with psychotic features, or Bipolar I in the past 24 months. Diagnosis of active substance dependence in the past 12 months or substance abuse in the last 6 months
* an immediate risk of suicide, requiring hospitalization or urgent evaluation
* clinician assessment that participation in the study could have an adverse impact on the patient or his/her partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2010-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia T. Valenstein, MD AB, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (4):
- United States (4):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Medical Center, Battle Creek, Battle Creek, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan
  - Aleda E. Lutz VA Medical Center, Saginaw, Michigan

REFERENCES:
- [Background] Pfeiffer PN, Heisler M, Piette JD, Rogers MA, Valenstein M. Efficacy of peer support interventions for depression: a meta-analysis. Gen Hosp Psychiatry. 2011 Jan-Feb;33(1):29-36. doi: 10.1016/j.genhosppsych.2010.10.002. Epub 2010 Nov 13. PMID 21353125
- [Result] Pfeiffer PN, Brandfon S, Garcia E, Duffy S, Ganoczy D, Myra Kim H, Valenstein M. Predictors of suicidal ideation among depressed Veterans and the interpersonal theory of suicide. J Affect Disord. 2014 Jan;152-154:277-81. doi: 10.1016/j.jad.2013.09.025. Epub 2013 Oct 4. PMID 24135507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a total of 15 VA mental health clinics, located within four VA Healthcare Systems and their affiliated Community Based Outpatient Centers.
Groups:
- Enhanced Usual Care: Enhanced Usual Care: Patients received a copy of the Depression Helpbook by Wayne Katon and bi-weekly study mailings with depression management tips.
- Telephone-based Peer Support: Telephone-based peer support: Patients received a) a peer-support manual that outlines self-management and recovery principles and provides peer discussion topics and b) access to a specialized telephone platform that permits free calls to their partners, ready access to mental health staff for back-up and advice on being effective partners, and recorded tips on depression management. They were asked to call their peer partner at least once a week for 24 weeks.
  Enhanced Usual Care: Patients received a copy of the Depression Helpbook by Wayne Katon and bi-weekly study mailings with depression management tips.
Period: Overall Study
Arm/Group | Enhanced Usual Care | Telephone-based Peer Support
Started | 243 | 200
Intervention Interruption | 0 | 56 (56 participants excluded from main analyses due to 2 mos interruption in study intervention)
Completed | 212 | 129
Not Completed | 31 | 71
Not completed — Lost to Follow-up | 25 | 9
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Death | 0 | 2
Not completed — Protocol Violation | 0 | 56

BASELINE CHARACTERISTICS:
Population: Fifty-six of the patients randomized to the telephone-based peer support intervention were excluded from main study analyses because of an unforeseen disruption in their 6-month intervention that was unrelated to patient characteristics.
Groups:
- Enhanced Usual Care: Patients in the enhanced usual care arm received their usual mental health care, a copy of the Depression Helpbook by Wayne Katon and bi-weekly study mailings with depression management tips.
  Enhanced Usual Care: Patients received a copy of the Depression Helpbook by Wayne Katon and bi-weekly study mailings with depression management tips.
- Telephone-based Peer Support: Participants used an IVR telephone system for mutual peer support over a 6-month period of time. Additionally, participants will received a copy of the Depression Helpbook by Wayne Katon and bi-weekly study mailings with depression management tips.
  Telephone-based peer support: Patients received a) a peer-support manual that outlines self-management and recovery principles and provides peer discussion topics and b) access to a specialized telephone platform that permits free calls to their partners, ready access to mental health staff for back-up and advice on being effective partners, and recorded tips on depression management. They were asked to call their peer partner at least once a week for 24 weeks.
  Enhanced Usual Care: Patients received a copy of the Depression Helpbook by Wayne Katon and bi-weekly study mailings with depression management tips.
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | Telephone-based Peer Support | Total
Number analyzed (Participants) | 243 | 144 | 387
Age, Customized [Number; unit: participants]
  18-44 years | 48 | 25 | 73
  45-64 years | 161 | 91 | 252
  > 65 years | 34 | 28 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 27 | 74
  Male | 196 | 117 | 313

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Status-Mental Health (MCS) Over 12 Month Period
Description: The Veterans Rand 36 Item Health Survey (VR-36) mental health component score (MCS) and physical health component score (PCS) were used as measures of functional status. The MCS and PCS have a mean of 50 and standard deviation of 10, with higher scores indicating better health.
Time Frame: Change over study period
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care | Telephone-based Peer Support
Number analyzed (Participants) | 240 | 137
units on a scale
  Baseline | 32.71 (9.91) | 33.72 (10.97)
  3-month | 34.77 (11.59) | 36.58 (11.23)
  6-month | 36.6 (11.48) | 37.52 (11.65)
  12-month | 36.99 (11.00) | 37.24 (11.14)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Telephone-based Peer Support; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = 0.22, 95% CI 2-sided [-1.57 to 2.01]

2. Primary Outcome: Change in Functional Status-Physical Health (PCS) Over 12 Month Period
Description: as for outcome 1
Time Frame: Change over study period
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care | Telephone-based Peer Support
Number analyzed (Participants) | 240 | 137
units on a scale
  Baseline | 36.63 (10.64) | 34.62 (10.44)
  3-month | 37.68 (11.10) | 35.14 (11.18)
  6-month | 36.91 (10.89) | 34.64 (11.31)
  12-month | 36.72 (11.16) | 35.48 (11.13)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Telephone-based Peer Support; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -0.39, 95% CI 2-sided [-2.03 to 1.24]

3. Primary Outcome: Quality of Life
Description: The 14-item Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF), which has good reliability and has been used in multiple depression studies, was used to assess quality of life. Responses are scored on a 5-point scale ('not at all or never' to 'frequently or all the time'), where higher scores indicate better enjoyment and satisfaction with life (possible range 14-70).
Time Frame: Change over study period
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care | Telephone-based Peer Support
Number analyzed (Participants) | 242 | 139
units on a scale
  Baseline | 38.80 (8.74) | 38.82 (9.22)
  3-Month | 41.14 (9.07) | 41.75 (9.42)
  6-Month | 41.89 (9.76) | 42.55 (9.66)
  12-month | 42.69 (9.97) | 42.55 (9.55)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Telephone-based Peer Support; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = 0.81, 95% CI 2-sided [-0.93 to 2.55]

4. Primary Outcome: Depression Symptoms
Description: The 21-item Beck Depression Inventory-2nd Edition (BDI-II) was used to assess depressive symptoms. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Change over study period
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care | Telephone-based Peer Support
Number analyzed (Participants) | 243 | 144
units on a scale
  Baseline | 25.60 (10.29) | 25.16 (11.34)
  3-Month | 20.77 (11.72) | 19.51 (11.23)
  6-month | 18.86 (11.63) | 18.17 (12.29)
  12-month | 17.82 (11.73) | 17.15 (10.86)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Telephone-based Peer Support; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -.039, 95% CI 2-sided [-2.66 to 1.89]

5. Primary Outcome: Recovery Orientation
Description: The 30-item Mental Health Recovery Measure (MHRM) was used to assess recovery orientation. The MHRM has been fielded among diverse populations and has a high level of internal consistency (Cronbach's α =.93) and shows change following engagement in recovery oriented treatments. The MHRM is scored using a 5 point Likert Scale (0 to 4) for each item, yielding a theoretical range from 0 - 120 for Total Score. Higher scores correspond to a higher self-reported level of mental health recovery.
Time Frame: Change over study period
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care | Telephone-based Peer Support
Number analyzed (Participants) | 239 | 138
units on a scale
  Baseline | 64.23 (18.89) | 64.10 (18.73)
  3-Month | 67.37 (19.98) | 68.47 (19.47)
  6-month | 71.25 (19.51) | 70.50 (20.08)
  12-month | 73.06 (19.82) | 69.81 (18.66)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Telephone-based Peer Support; Test type: Superiority or Other; Slope = -.08, 95% CI 2-sided [-3.31 to 3.16]

ADVERSE EVENTS:
Time Frame: Time frame was March 2010-October 2013 for a total of 3 years and 7 months.
Arm/Group | Enhanced Usual Care | Telephone-based Peer Support
Serious Adverse Events (participants affected / at risk) | 5/243 | 2/144
Other Adverse Events (participants affected / at risk) | 0/243 | 0/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enhanced Usual Care (N=243) | Telephone-based Peer Support (N=144)
Death (Cardiac disorders) | 0 | 2
Inpatient Psychiatric Hospitalization (Psychiatric disorders) | 5 | 0

LIMITATIONS AND CAVEATS:
56 of the patients randomized to the telephone-based peer support intervention were excluded from main study analyses because of an unforeseen disruption in their 6-month intervention that was unrelated to patient characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes